CLINICAL TRIAL: NCT02241031
Title: Megakaryocytic Progenitor Cells for Prophylaxis and Treatment of Thrombocytopenia in Patients With Acute Leukemia Receiving Chemotherapy
Brief Title: Megakaryocytic Progenitor Cells for Prophylaxis and Treatment of Thrombocytopenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Southern Medical University, China (Other); Peking University People's Hospital (Other); Huazhong University of Science and Technology (Other); Sun Yat-sen University (Other); Academy Military Medical Science, China (Industry)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPs-AL-2014
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Hematological Diseases; Thrombocytopenia
Keywords: Megakaryocytic Progenitor Products; Hematological Diseases; Thrombocytopenia
MeSH Terms: conditions — Hematologic Diseases; Thrombocytopenia | interventions — Thrombopoietin; Interleukin-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPs (Experimental): MPs will be intravenously infused within 48 hours after chemotherapy. During the study period, patients can receive platelet infusion but can not receive platelet stimulating factors.
  Interventions: Biological: MPs
- Non-MPs (Active Comparator): Patients can receive platelet infusion but can not receive platelet stimulating factors.
  Interventions: Drug: thrombopoietin (TPO) and interleukin-11

INTERVENTIONS:
Biological: MPs — MPs are generated from cord blood using a combination of cytokines.
  Arms: MPs
Drug: thrombopoietin (TPO) and interleukin-11 — Platelet stimulating factors include thrombopoietin (TPO) and interleukin-11 and so on.
  Arms: Non-MPs

SUMMARY:
The purpose of this study is to evaluate the efficacy of ex vivo generated megakaryocytic progenitor cells (MPs) in prophylaxis and treatment of thrombocytopenia caused by chemotherapy in patients with acute leukemia (AL).

DETAILED DESCRIPTION:
Thrombocytopenia is a common and potentially fatal complication of chemotherapy and hematopoietic stem cell transplantation. Owing to the short storage time and increased demand of platelets from unrelated donors, a constant shortage in the supply of platelets has become an important medical and society challenge. Therefore, investigation of alternative sources of platelets would be beneficial.

Hematopoietic stem cells (HSCs) can be used to generate functional megakaryocytic progenitors (MPs), megakaryocytes, and platelets on a large scale. Functional MPs and platelets have successfully been produced in vitro from CD34+ hematopoietic cells from bone marrow, cord blood, and peripheral blood. Several studies have reported that transplantation of in vitro auto-producing MPs can promote platelet recovery after high-dose therapy and HSC transplantation.

Umbilical cord blood is an abundant source of HSCs. In vitro large scale production of MPs from cord blood could represent an effective platelet substitute. Theoretically, the additional transplantation of ex vivo generated progenitor and post-progenitor cells might lead to the production of sufficient numbers of mature functional cells within a few days after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age：14-65 years
* achieve complete remission of acute leukemia
* the first course of consolidation chemotherapy
* ECOG grades 0 or 1
* expected survival time ≥ three months
* Subjects (or their legally acceptable representatives) must have signed an informed consent document.

Exclusion Criteria:

* cardiac dysfunction (particularly congestive heart failure), hepatic abnormalities (bilirubin ≥ 3 mg/dL, aminotransferase> 2 times the upper limit of normal), renal dysfunction (creatinine clearance rate < 30 mL/min)
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Platelet recovery after infusion of MPs | 3 months
  Platelet recovery after infusion of MPs includes the time from infusion to platelet count≥20×10^9/L,50×10^9/L,100×10^9/L.

SECONDARY OUTCOMES:
frequency of platelet infusion | 3 months
incidence of acute toxicity | 3 month
  Acute toxicity mainly involves the heart,live and kidney.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Xi J, Zhu H, Liu D, Nan X, Zheng W, Liu K, Shi W, Chen L, Lv Y, Yan F, Li Y, Xie X, Wang Y, Yue W, Xu X, Wei X, Zhu J, Huang X, Pei X. Infusion of megakaryocytic progenitor products generated from cord blood hematopoietic stem/progenitor cells: results of the phase 1 study. PLoS One. 2013;8(2):e54941. doi: 10.1371/journal.pone.0054941. Epub 2013 Feb 4. PMID 23390507